CLINICAL TRIAL: NCT05471557
Title: Effects of Acute Pain on Motor Learning in Young vs Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susanne M Morton, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1786370-1.1; R01AG071585 (NIH)
Record Dates: First submitted 2022-07-17; First posted 2022-07-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Aging; Pain, Acute; Cognitive Decline; Motor Activity
Keywords: Acute pain; Adults; Cognition; Elderly; Learning; Memory; Pain; Cognitive ability; Motor learning; Young adults; Older Adults; Gait; Locomotion; Walking; Motor Consolidation
MeSH Terms: conditions — Acute Pain; Cognitive Dysfunction; Motor Activity; Pain

STUDY DESIGN:
Masking Description: Application of pain or no stimulus cannot be masked from participants, nor from outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Stimulus (Experimental): Capsaicin combined with heat applied to intact skin
  Interventions: Procedure: pain delivery
- No Stimulus (No Intervention): Nothing applied to skin

INTERVENTIONS:
Procedure: pain delivery — Experimental pain paradigm delivered that is short-term and painful but not harmful.
  Arms: Pain Stimulus

SUMMARY:
To date, the effects of pain on motor learning have not been thoroughly investigated, particularly in older adults. Broadly, the purpose of this research is to investigate the impact of acute pain on locomotor learning and its retention in older adults. The investigators hypothesize that acute pain impairs retention of locomotor learning in young and older adults and that in older adults, these deficits are worsened and are related to the degree of normal age-related cognitive decline.

ELIGIBILITY:
Abbreviations: YA= young adult; OA= older adult; HR= heart rate, bpm= beats per minute; BP= blood pressure; ADD= attention deficit disorder; ADHD= attention deficit hyperactivity disorder; MoCA= Montreal Cognitive Assessment; GAD-7= Generalized Anxiety Disorder 7 Scale; PHQ-2, PHQ-9= Patient Health Questionnaire-2 and -9.

Inclusion Criteria:

1. 18-35 (YA group only) or 55-85 (OA group only) years old
2. Sex-matched to a participant in the OA group (YA group only)
3. Self-identifying as generally medically healthy
4. Able to read, write and speak English
5. Able to provide informed consent and attend all testing sessions
6. Willing to undergo the experimental pain or non-painful electrical stimulation, if selected

Exclusion Criteria:

1. Resting HR < 50 or > 100 bpm
2. Resting BP < 90/60 or > 140/95 mmHg (YA group only) or > 165/95 (OA group only)
3. Any history or current mental health condition, learning/developmental disability or cognitive impairment, including severe untreated ADD/ADHD, severe untreated anxiety, severe untreated depression, autism spectrum disorder, insomnia, mild cognitive impairment, etc.
4. Score on the MoCA <23
5. Score on the GAD-7 ≥ 10
6. Score on the PHQ-2 ≥ 2 and score on the PHQ-9 ≥ 10
7. Any current (within last 3 month) or chronic medical conditions, including any musculoskeletal, cardiovascular, endocrine, pulmonary, metabolic, psychiatric or neurological diagnosis that (for OA group only) affects activities of daily living or would confound testing or place the subject at risk by participating, such as a significant cardiovascular condition or event (e.g., heart attack < 3 months ago, uncontrolled atrial fibrillation, uncontrolled angina, or congestive heart failure, chronic obstructive pulmonary disorder, peripheral vascular disease)
8. Any impaired sensation or weakness in either lower extremity or in the area targeted for the stimulus
9. History of serious concussion or head injury, defined as a loss of consciousness for > 5 minutes and/or requiring medical treatment, or > 2 concussions over the lifespan
10. Any history of acute or chronic problems with balance, any dizziness, or > 1 fall in the last 12 months
11. Taking 4 or more medications (YA group only)
12. Currently or regularly using any analgesic medications, over-the-counter remedies, or any other treatment for the purposes of pain relief (i.e., baby aspirin for heart health permitted, etc.)
13. Any current or chronic pain condition during the last year, located anywhere in the body with a (OA group only) pain intensity of > 2/10
14. Allergy to capsaicin or hot peppers
15. Any skin lesion, breakage or irritation in the area targeted for the painful stimulus
16. Skin sensitivity to soaps/creams/perfumes or to heat
17. Poor circulation in the area targeted for the painful stimulus
18. Prior participation in a locomotor learning study in this lab within the last 2 years or prior participation in a study in this lab that included the cognitive testing battery within the last 2 years.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Motor Retention Magnitude | 24 hours post learning (day 2)
  degree to which the learned locomotor pattern has been remembered (in step length % change, normalized to the amount learned from day 1)
Motor Learning Magnitude | immediately after learning (day 1)
  degree to which the new locomotor pattern has been acquired (in step length % change)
Digit Span Backward Test | the change between baseline and during application of intervention
  number of digits (numbers) that can be repeated back in the reverse order from which they were presented
Digit Span Forward Test | the change between baseline and during application of intervention
  number of digits (numbers) that can be repeated back in the same order as they were presented

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Morton, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

REFERENCES:
- [Background] Patel KV, Guralnik JM, Dansie EJ, Turk DC. Prevalence and impact of pain among older adults in the United States: findings from the 2011 National Health and Aging Trends Study. Pain. 2013 Dec;154(12):2649-2657. doi: 10.1016/j.pain.2013.07.029. PMID 24287107
- [Background] Whitlock EL, Diaz-Ramirez LG, Glymour MM, Boscardin WJ, Covinsky KE, Smith AK. Association Between Persistent Pain and Memory Decline and Dementia in a Longitudinal Cohort of Elders. JAMA Intern Med. 2017 Aug 1;177(8):1146-1153. doi: 10.1001/jamainternmed.2017.1622. PMID 28586818
- [Background] Higgins DM, Martin AM, Baker DG, Vasterling JJ, Risbrough V. The Relationship Between Chronic Pain and Neurocognitive Function: A Systematic Review. Clin J Pain. 2018 Mar;34(3):262-275. doi: 10.1097/AJP.0000000000000536. PMID 28719507
- [Background] Institute of Medicine (US) Committee on Advancing Pain Research, Care, and Education. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK91497/ PMID 22553896
- [Background] van der Leeuw G, Leveille SG, Dong Z, Shi L, Habtemariam D, Milberg W, Hausdorff JM, Grande L, Gagnon P, McLean RR, Bean JF. Chronic Pain and Attention in Older Community-Dwelling Adults. J Am Geriatr Soc. 2018 Jul;66(7):1318-1324. doi: 10.1111/jgs.15413. Epub 2018 Jun 6. PMID 29876923